CLINICAL TRIAL: NCT05303870
Title: Exploring the Transferability of Improving Access to Psychological Therapies (IAPT) to a General Hospital Emergency Inpatient Ward
Brief Title: Impact of Psychological Therapies on Emergency Medical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Suffolk and North Essex NHS Foundation Trust (Other)
Collaborators: University of Essex (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/024
Record Dates: First submitted 2022-02-21; First posted 2022-03-31 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Mental Health Disorder; Mental Disorder; Mental Health Wellness 1
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IAPT (Experimental)
  Interventions: Other: Improving access to psychological therapies (IAPT)

INTERVENTIONS:
Other: Improving access to psychological therapies (IAPT) — IAPT services provide evidence-based treatments for people with depression and anxiety disorders, and comorbid long-term physical health conditions or medically unexplained symptoms. IAPT services are characterised by three key principles:
  1. Evidence-Based psychological therapies at the appropriate dose: NICE recommended therapies matched to the mental health problem, at the intensity and duration designed to optimise outcomes.
  2. Appropriately trained and supervised workforce.
  3. Routine outcome monitoring.

SUMMARY:
Prevalence of anxiety and depression in the general population is known, but is under researched in the acute hospital setting and there is little evidence on the prevalence of anxiety and depression within the emergency medical admission population. A potential intervention for treating such mental health prevalence would be in the form of IAPT methodology which has been utilised in other parts of the NHS demonstrating good outcomes. Therefore, this feasibility study will explore the utility of IAPT in the acute setting.

This study will explore the prevalence of anxiety and depression in the emergency medical population within medical inpatient wards , utilising the assessment tools adopted by the IAPT services and explained in detail below.

The study will explore a) feasibility of introducing psychological intervention to an emergency medical ward and b) provide preliminary data on the outcome of this intervention on hospital length of stay and readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Ipswich Hospital into a ward that cares for patients who are medical emergencies.
* Patients who score 3 or higher on one or both of the GAD 2 and PHQ 2.
* Patients that have capacity to consent.
* Over 18 years old.
* Ability to speak and read in English as the study will not have the resources to employ interpreters or to get documentation translated.
* Participants that are not deemed suicidal via screening and medical and nurse assessment.

Exclusion Criteria:

* Patients not receiving care on a ward caring for medical emergencies.
* Patients under the age of 18 years old.
* Patients scoring < 3 on both GAD 2 and PHQ 2.
* Patients who do not have capacity to consent.
* Participants that are suicidal as via screening and medical and nurse assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with moderate or severe anxiety | Up to 6 months
  How many participants enrol in to the study, that are eligible to participate.

SECONDARY OUTCOMES:
IAPT views | Up to 6 months
  Thematic analysis of in depth interviews on staff and patients regarding the IAPT intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- East Suffolk and North Essex NHS Foundation Trust, Ipswich, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided